CLINICAL TRIAL: NCT06622980
Title: The Effect of an Ergonomic Educational Intervention on Laparoscopic Surgeons' Ergonomic Risk Scores
Brief Title: The Effect of an Ergonomic Educational Intervention on Laparoscopic Surgeons' Ergonomic Risk Scores (ErgoEd)
Acronym: ErgoEd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MKUH-RD-027; 332452 (Other: IRAS)
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Surgery, Laparoscopic
Keywords: laparoscopic surgery; ergonomics; ergonomic education; Ergonomic Risk Score; REBA
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Single arm pre-post study with the educational intervention taking place outside of the clinical setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laparoscopic surgeons (Experimental): Laparoscopic surgeons from any surgical subspecialty
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The educational intervention will take the form of a video explaining both general ergonomic principles and specific advice for laparoscopic surgeons. This video will be shown to surgeons at a time of their convenience and the research team will be available to answer any further questions at this time.
  The educational video will cover both ergonomics principles and specific advice for laparoscopic surgeons. The principles will be relevant to any situation, including those outside the medical field. The laparoscopic-specific section will include tips for optimisation of operating theatre set-up and advice on posture and body position. The video content will be reviewed by experts experienced in surgical ergonomics education to ensure it covers all useful information and is in line with best practice.

SUMMARY:
This study aims to determine whether education of surgeons can reduce the physical strain of performing surgery. Laparoscopic surgery is known to be beneficial for patients but can cause both short- and long-term musculoskeletal injuries for the surgeons who perform it. The purpose of the study is to investigate whether the physical risks to surgeons can be reduced by educating them on how to best set up the operating theatre and equipment, and how to optimise their posture and position whilst operating.

DETAILED DESCRIPTION:
This study has been designed to assess whether receiving education in ergonomic principles can lower surgeons' ergonomic risk scores when performing laparoscopic surgery. The study will recruit surgeons who regularly perform laparoscopic surgery, with no stipulations on surgeon speciality. All surgeons will be required to have completed at least 20 laparoscopic cases beforehand.

The primary outcome will be assessed intraoperatively, with additional questionnaire data collected immediately postoperatively. Assessment of ergonomics (REBA score) will be done from still photographs that focus on the operating surgeon, although other team members may be visible in the background. Photographs will be analysed postoperatively by the research team and an overall REBA score calculated for each surgeon.

Other secondary outcomes will be assessed via a questionnaire. After each operation surgeons will complete a subjective cognitive and physical strain questionnaire based on the NASA-TLX and SURG-TLX scales, which are both widely used and validated tools. Additional questions have been added in order to provide data for the development of a new subjective physical strain questionnaire based on pooled data from several surgical ergonomics trials.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic surgeon from any surgical subspecialty
* Can commit sufficient time to ergonomic training

Exclusion Criteria:

• Training grade more junior than a registrar

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Rapid Entire Body Assessment (REBA) score | (1) operating list before the intervention - no specified time frame, (2) operating list 1 week after the intervention, (3) operating list 4-6 weeks after the intervention.
  To assess whether receiving education on ergonomics can reduce laparoscopic surgeons' ergonomic risk (REBA) scores whilst operating.
  The risk score is calculated post hoc from photographs taken every 1-minute for the duration of operating for each 3 observed operating lists. One operating list may include more than one operation.

SECONDARY OUTCOMES:
Cognitive and physical strain score | Questionnaire taken immediately at the end of each observed operation.
  To compare surgeons' subjective experience of pain and discomfort intraoperatively.
  This is a modified questionnaire including items from Hart and Staveland's NASA Task Load Index (NASA-TLX) and Wilson et al. the surgery task load index (SURG-TLX).
  Higher scores indicate higher cognitive and physical strain.
Feedback questionnaire on educational intervention | Completed once immediately after the final (third) observed operating list (4-6 weeks after the intervention)).
  To gain feedback on the design of the educational intervention.
Ergonomic knowledge questionnaire | Assessed at baseline - immediately after consent - but prior to first observed operating list (no timeframe specified), and again immediately after final (third) observed operating list (4-6 weeks after the intervention).
  To assess whether surgeons' theoretical knowledge of ergonomic principles can be improved
Acceptability of recruitment and study retention | at the end of the trial (last surgeon's third operating list/4-6 weeks after the last recruited surgeon has received the intervention)
  This measurement is part of the feasibility of a future larger-scale study. This is measured through an assessment of how many participants decline to participate or withdraw from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Barrie Keeler, Principal Investigator — Milton Keynes University Hospital
Locations (1):
- Milton Keynes University Hospital, Milton Keynes, Buckinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
R&D will evaluate requests on a case-by-case basis.